CLINICAL TRIAL: NCT01794338
Title: A Randomized, Prospective, Double Blind Clinical Trial of Non-cross-linked Porcine Dermis vs. Bioabsorbable Synthetic Mesh for the Repair of Abdominal Wall Defects in At-risk Patients
Brief Title: The Use of Biologic Mesh vs Bioabsorbable Mesh During Ventral Hernia Repair in At-risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of incorporation with patients
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-12-02A
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-04

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bio-A Arm (Experimental): Patients will receive underlay mesh tissue reinforcement followed by standard fascial closure with #1 PDS. As described by Dr. Stoppa10-12, the mesh will be secured via abdominal wall sutures. Additional full thickness sutures will be placed every 8 cm circumferentially. After securing the mesh in place, #1 PDS sutures will be used to close the fascia in a running fashion with 1.5-2 cm "bites" from the fascial edge and a 1cm "walk" between stitches. Skin will be closed with staples or monofilament suture according to surgeon preference. Drains will be placed on the mesh in each case, and one or two drains will be placed in the subcutaneous tissues at the discretion of the surgeon depending on the amount of subcutaneous tissue dissected.
  Interventions: Device: Bio-A Arm
- Strattice Arm (Active Comparator): Patients will receive underlay mesh tissue reinforcement followed by standard fascial closure with #1 PDS. As described by Dr. Stoppa10-12, the mesh will be secured via abdominal wall sutures. Additional full thickness sutures will be placed every 8 cm circumferentially. After securing the mesh in place, #1 PDS sutures will be used to close the fascia in a running fashion with 1.5-2 cm "bites" from the fascial edge and a 1cm "walk" between stitches. Skin will be closed with staples or monofilament suture according to surgeon preference. Drains will be placed on the mesh in each case, and one or two drains will be placed in the subcutaneous tissues at the discretion of the surgeon depending on the amount of subcutaneous tissue dissected..
  Interventions: Device: Strattice Arm

INTERVENTIONS:
Device: Strattice Arm — Biologic mesh to be placed during hernia repair surgery
  Arms: Strattice Arm
Device: Bio-A Arm — Bioabsorbable mesh to be placed during hernia repair surgery
  Arms: Bio-A Arm

SUMMARY:
This study evaluates the outcomes of patients who have been treated with Strattice or Gore Bio-A mesh for the repair of complicated abdominal wall hernias. The purpose of this study is to collect information and evaluate the outcome of your surgery. Synthetic (man made) mesh has been shown to provide durable long-term outcomes; however, this type of mesh should not be used in patients at risk of developing an infection. Therefore, to address the challenge of finding an artificial strengthening material to repair complicated hernias in patients that could potentially develop surgical infection, two types of non-permanent materials have been developed, including biologics and bioabsorbables. Biologic mesh is made of living tissue and bioabsorbable mesh is made of synthetic material that is gradually absorbed by the body over time. The purpose of this study is to allow surgeons to compare the postoperative course of patients associated with these two mesh types to decide which material will improve the outcomes of their patients with complicated abdominal wall defects. To date there is no evidence to suggest that either mesh type is superior or safer than the other.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the outcomes of patients implanted with Strattice® (LifeCell Corporation, Branchburg, NJ, USA) and Gore® Bio-A® (W. L. Gore & Associates, Inc., Newark, DE, USA) for the repair of abdominal wall defects in at-risk patients. Primary endpoints of the study will include hernia recurrence, duration of postoperative drains, the incidence of systemic and wound-related complications, the need for percutaneous intervention or reoperation and quality- of-life with 3 years of follow-up. The study will be prospective and randomized, and the evaluator and patient will be blinded as to the type of mesh implanted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Grade II or III ventral hernia according to Ventral Hernia Working Group (VHWG)
* Pre-operative informed consent is obtainable

Exclusion Criteria:

* Return to the operating room within the next 1 year for additional open abdominal surgery is anticipated
* Absence of fascial defect or fascial defect less than 3 cm in greatest dimension
* Presence of previously place mesh (synthetic or biologic) at the site of surgery, which will not be completely removed and will, in part or whole, remain at the site of implantation of the study mesh
* Concurrent placement of another mesh (synthetic or biologic) at the site where the study mesh is placed
* Grade IV ventral hernia according to VHWG system
* ASA score IV or above
* Any disease or condition along with the surgeon's clinical judgment that contraindicates the use of either study mesh
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant T Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bio-A Arm | Strattice Arm
Started | 8 | 9
Screen Failure | 3 | 3
1 Month Follow Up | 6 | 9
6 Month Follow Up | 0 | 0
12 Month Follow Up | 0 | 0
24 Month Follow Up | 0 | 0
36 Month Follow Up | 0 | 0
Completed | 0 | 0
Not Completed | 8 | 9
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 6 | 9

BASELINE CHARACTERISTICS:
Population: The study was terminated before reaching full enrollment needed for analysis. Per https://clinicaltrials.gov/ct2/manage-recs/faq#terminated (accessed on 1.31.2019) we have indicated 0 for each study arm. Numbers were updated to reflect participants at the time of study termination. Baseline data were NOT COLLECTED
Groups:
- Total: Total of all reporting groups
Arm/Group | Bio-A Arm | Strattice Arm | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — Population: This research project enrolled 28 subjects, 9 subjects were excluded due to various factors, 2 subjects are deceased due to non-study related factors and 15 subjects were lost to follow-up. The study was terminated because of lack of active subjects and low recruitment. No analyses were performed as the study was terminated due to lack of enrollment and patients lost to follow up. As a result of the lack of enrollment and patients lost to follow up, data were not collected.
Sex/Gender, Customized — Population: No analyses were performed as the study was terminated due to lack of enrollment and patients lost to follow up. As a result of the lack of enrollment and patients lost to follow up, data were not collected.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hernia Recurrence
Description: Patients will undergo post-operative follow-up at 1 month, 6 months, and yearly for 3 years. Patients will receive reminders of their follow-up visits before each time period. At each visit, patients will be asked to fill out a short questionnaire (Form A and Form B) that will aid in assessing and documenting postoperative symptoms and quality of life. During each follow-up visit a board certified or board eligible surgeon, who is blinded with regard to the group assignment, will perform a physical examination to assess for the presence of a recurrent hernia, eventration and other findings detailed on Form C. Any signs of wound complications will be noted, including seroma formation, erythema, drainage, break in the skin, purulence or tenderness to palpation. If a recurrent hernia defect is identified on the physical examination, imaging studies will be performed as indicated. Once a hernia defect is found, further management options will be discussed with the patient.
Time Frame: 3 years
Population: The study was terminated before reaching full enrollment needed for analysis. Per https://clinicaltrials.gov/ct2/manage-recs/faq#terminated (accessed on 1.31.2019) we have indicated 0 for each study arm. No analyses were performed as the study was terminated due to lack of enrollment and patients lost to follow up and therefore no data was able to be collected for analysis.
Arm/Group | Bio-A Arm | Strattice Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event will be reported to the IRB within 48 hours of event occurrence. Participants were followed until study completion. Participants would be followed for 1 year however all eligible participants were lost to follow up.
Description: Definitions do not differ.
Groups:
- Bio-A Arm: bioabsorbable mesh
- Strattice Arm: common biologic mesh originating from porcine dermal matrix
Arm/Group | Bio-A Arm | Strattice Arm
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT01794338/Prot_SAP_000.pdf